CLINICAL TRIAL: NCT04845698
Title: Application of i-Dashboard for Multi-disciplinary Rounds in Surgical Intensive Care Units
Brief Title: i-Dashboard for Multi-disciplinary Rounds in SICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chao-Han Lai, MD, PhD, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: B-ER-110-040
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Workflow; Communication; Quality of Health Care
Keywords: Electronic Health Records; User-Computer Interface; Intensive Care Units; Patient Care Team; Teaching Rounds
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: A cluster randomized trial was conducted in two surgical intensive care units (ICUs) of the hospital. For each two-week period of the trial, participating ICUs (cluster) were assigned to multi-disciplinary rounds with i-Dashboard (intervention) or without i-Dashboard (control). In other words, the two ICUs were randomly assigned to multi-disciplinary rounds with i-Dashboard during the first two weeks, without i-Dashboard during the second two weeks, and with i-Dashboard during the third two weeks or vice versa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With i-Dashboard (Experimental): Multi-disciplinary rounds are conducted with the assistance of i-Dashboard.
  Interventions: Device: i-Dashboard
- Without i-Dashboard (No Intervention): Multi-disciplinary rounds are conducted without the assistance of i-Dashboard. The team members collect data using standard electronic medical records.

INTERVENTIONS:
Device: i-Dashboard — i-Dashboard is a team-designed, patient-centered electronic medical record viewer, which retrieves data from multiple databases and provides a quick representation of essential metrics for each patient.
  Arms: With i-Dashboard

SUMMARY:
Background: Information overload is a common problem in intensive care units. A display tool that facilitates retrieval of crucial clinical information from electronic medical records has excellent potential to attenuate information overload and benefit workflow.

Study hypothesis: In this project, we aimed to evaluate the efficacy and clinical satisfaction of a team-designed, patient-centered electronic medical record viewer, i-Dashboard, to facilitate multi-disciplinary rounds in our surgical intensive care units.

DETAILED DESCRIPTION:
Background: More than 5.7 million people are admitted into intensive Care Units (ICUs) in the United States each year. The ICU level of care that helps people with a life-threatening illness is provided by a multi-disciplinary team of specially-trained healthcare providers. These patients require more frequent assessment compared to those who do not need critical care. Essential parameters in the ICU settings include, but not limit to, vital sign monitoring, laboratory data, ventilator settings and vasoactive drugs. Therefore, information overload is a common problem in ICUs. Caring for ICU patients generates approximately 1200 data points per patient per day. The use of electronic medical records (EMRs) increases the data accuracy compared to handwritten notes. An effective management strategy for patient information in ICUs may be needed for clinicians to avoid being overwhelmed by data overload.

Data overload in ICUs may result in communication failures, possibly in association with worse patient outcomes. A delay between condition onsets and the beginning of therapeutic interventions may dramatically impact the prognosis of patients with sepsis or cardiopulmonary emergencies. Although EMR use has been increasingly adopted worldwide, whether EMRs are being used effectively and efficiently to enhance clinical workflow in ICUs remains a question. A large cross-sectional study of primary care practitioners have investigated the predictors of missed test results in the setting of EMR alerts. Of the 2590 responders, 86.9% perceived the quantity of alerts they received to be excessive, 69.6% reported receiving more alerts than they could effectively manage (a marker of information overload), 55.6% reported that the current EMR notification system made it possible for practitioners to miss test results, and 29.8% reported having personally missed test results that led to care delays. These results suggested that primary care practitioners using comprehensive EMRs are vulnerable to information overload, leading them to miss important information. To address the nature of the high volume of metrics monitored and the urgent responses to patients' condition changes in ICUs, a display tool that facilitates retrieval of crucial clinical information has excellent potential to attenuate information overload and benefit workflow.

Visualization transforms data into visual representations, making the cognitive processing of data more effective and efficient. The use of visualization techniques in the clinical setting provides an overview to improve display and recognition of patients' conditions, potentially reducing cognitive overload among specially-trained healthcare providers. A dashboard is a data-driven clinical decision support tool capable of retrieving data from multiple databases and providing a quick representation of key metrics for each patient. The utility of a dashboard comes from its ability to provide a concise overview of crucial information. In addition to being designed based on user experiences, a dashboard for clinical use should be designed based on several proposed principles, including 1) one view should contain single patient data, 2) data should be summarized or titled for overview and details should be given on-demand, 3) data should be displayed in time-series, 4) data should be categorized by primary type, and 5) more data should be displayed at the same time. While being applied to the ICU settings, a dashboard may allow healthcare providers in a multi-disciplinary team to identify patients' active problems that need prompt interventions.

Hypothesis and Specific Aims: The implementation of multi-disciplinary rounds in ICUs exhibits a positive effect on both patient care outcome and staff satisfaction with team dynamics. In Taiwan, multi-disciplinary ICU rounds have been an important item to be evaluated in hospital accreditation. The study participants include ICU healthcare providers, i.e. physicians, nurse practitioners, nurses, respiratory therapists, pharmacists and dietitians. In this project, we aimed to evaluate the efficacy and clinical satisfaction of a team-designed, patient-centered electronic medical record viewer, i-Dashboard, to facilitate multi-disciplinary rounds in our surgical intensive care units. To achieve these research goals the applicant proposed studies with the following specific aims:

1. The use of i-Dashboard reduces time spent on pre-round data gathering.
2. The use of i-Dashboard increases communication accuracy during multi-disciplinary ICU rounds, including vital signs, catheters, laboratory data, medications, input/output balance and warnings on redline values.
3. The use of i-Dashboard enhances recommendations actively made by multi-disciplinary team members, including respiratory therapists, pharmacists and dietitians.
4. The use of i-Dashboard enhances healthcare provider satisfaction, as evaluated by questionnaires modified from previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted into the two surgical intensive care units for more than 7 days

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-18 (Actual)

PRIMARY OUTCOMES:
Time spent on pre-round data gathering (minutes) | 3 hours
  Pre-round data gathering for multi-disciplinary rounds in ICUs is usually time-consuming. i-Dashboard, the team-designed display tool that facilitates retrieval of crucial clinical information from electronic medical records, is available on every computer screen in the ICU. We aim to evaluate whether i-Dashboard might help reduce time spent on pre-round data gathering for each patient evaluated during multi-disciplinary ICU rounds.
Communication accuracy during multi-disciplinary ICU rounds (number of data misrepresentation) | 3 hours
  Communication during multi-disciplinary ICU rounds relies primarily on handwritten notes. Based on the literature review, data misrepresentation commonly occurs during ICU rounds, and thus communication accuracy is highly questionable. i-Dashboard, the team-designed display tool, is designed to post the information on a 55-inch screen. We aim to evaluate whether i-Dashboard might help improve communication accuracy during multi-disciplinary ICU rounds.

SECONDARY OUTCOMES:
Enhancement of care quality and patient safety during multi-disciplinary ICU rounds (number of recommendations from multi-disciplinary team members) | 3 hours
  Multi-disciplinary team members in ICU (i.e., respiratory therapists, pharmacists and dietitians) provide their recommendations based on patients' condition and their own knowledge and expertise. These recommendations might be adopted by other team members. i-Dashboard, the display tool reporting the information on a large screen, might keep the multi-disciplinary team on the same page and help the members perceive patients' condition and other members' considerations. Thus, persuasive recommendations that enhance care quality and patient safety might be increased during multi-disciplinary rounds.
Healthcare provider satisfaction (questionnaire) | 3 months
  i-Dashboard might facilitate the multi-disciplinary ICU rounds and thus enhance healthcare provider satisfaction. The healthcare provider satisfaction will be evaluated by questionnaires modified from previous studies.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Han Lai, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital; Meng-Ru Shen, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, R.o.c, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pickering BW, Dong Y, Ahmed A, Giri J, Kilickaya O, Gupta A, Gajic O, Herasevich V. The implementation of clinician designed, human-centered electronic medical record viewer in the intensive care unit: a pilot step-wedge cluster randomized trial. Int J Med Inform. 2015 May;84(5):299-307. doi: 10.1016/j.ijmedinf.2015.01.017. Epub 2015 Jan 31. PMID 25683227
- [Background] Artis KA, Dyer E, Mohan V, Gold JA. Accuracy of Laboratory Data Communication on ICU Daily Rounds Using an Electronic Health Record. Crit Care Med. 2017 Feb;45(2):179-186. doi: 10.1097/CCM.0000000000002060. PMID 27655323
- [Background] Khairat SS, Dukkipati A, Lauria HA, Bice T, Travers D, Carson SS. The Impact of Visualization Dashboards on Quality of Care and Clinician Satisfaction: Integrative Literature Review. JMIR Hum Factors. 2018 May 31;5(2):e22. doi: 10.2196/humanfactors.9328. PMID 29853440
- [Derived] Lai CH, Li KW, Hu FW, Su PF, Hsu IL, Huang MH, Huang YT, Liu PY, Shen MR. Integration of an Intensive Care Unit Visualization Dashboard (i-Dashboard) as a Platform to Facilitate Multidisciplinary Rounds: Cluster-Randomized Controlled Trial. J Med Internet Res. 2022 May 13;24(5):e35981. doi: 10.2196/35981. PMID 35560107